CLINICAL TRIAL: NCT06625255
Title: Promoting Playfulness: Tier 1 Strength-based Parent Education Program to Promote Child and Family Resilience
Brief Title: Promoting Playfulness
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Florida Gulf Coast University (Other)
Collaborators: Yeshiva University (Other)
Responsible Party: Principal Investigator, Dr. Sarah Fabrizi, Associate Professor, Florida Gulf Coast University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Protocol ID # 2024-85
Record Dates: First submitted 2024-10-01; First posted 2024-10-03 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Developmental Delay (Disorder)
Keywords: play; playfulness; parent education
MeSH Terms: conditions — Developmental Disabilities

STUDY DESIGN:
Intervention Model Description: Flyers will be distributed, and participants will be able to contact the PI via email and use the QR code to complete the screening for eligibility. Eligibility screening will be conducted online by the prospective participant answering the following questions: (1) do you have a child aged 2 to 5? (b) do you speak and read English? and (c) can you attend two online sessions via Zoom where the content be provided via PowerPoint slides? Next, eligible participants will be asked to provide their email address and will then receive a link to complete the online consent procedure and pre-test through Qualtrics along with an assigned code to connect their pre-and-post data. The intervention group will begin when there are at least five eligible parents who consented. New enrolled parents will be waitlisted for two to three weeks after they completed the pre-program questionnaires, then after a two-week wait period they will be asked to complete the post-test Qualtrics survey 3.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention - Parent Education (Experimental): Parents will participate in 2, 45 minute virtual training sessions with information and question and anwsers. Each session will provide information about child development and parent advocacy and stressors. Play as the means for promoting healthy development will be emphasized.
  Interventions: Behavioral: Parent Education - Promoting Playfulness
- Waitlist control (No Intervention): Parents will have family life as usual with no education sessions.

INTERVENTIONS:
Behavioral: Parent Education - Promoting Playfulness — Parents will participate in 2, 45 minute parent education sessions promoting playfulness through information about child development, parent stressors, and parent advocacy.
  Arms: Intervention - Parent Education

SUMMARY:
Health inequalities, social isolation, and family adversity impact a child's development. Play is the context for child development in all areas. A parent's ability to support children at play while being playful contributes to their psychological adjustment. The proposed tier 1, strengths-based educational program for parents of children aged 2 to 5 years with and without disabilities combines elements of a play-based approach and tips on effective parenting to support children's development by equipping parents with knowledge and empowering them to become change agents in their children's lives.

DETAILED DESCRIPTION:
Parents will be recruited through a convenience sampling method to either an intervention group delivered online or a control waitlist group. Parents will be asked to complete a set of questionnaires online to assess the proposed programs effectiveness. Data analysis will explore between and within group differences in parental sense of competency, parental stress, child's behavior, and ability to support child's play. Qualitative data will be collected through online open-ended questions and sessions' transcript which will be analyzed to identify benefits. The project will produce tangible outcomes that will contribute to fostering the resilience of families with young children.

ELIGIBILITY:
Inclusion Criteria:

* Parent of a child aged 2 to 5 with no major disability (sensory, intellectual disability, neuromuscular disability).
* Can commit to participating in two online sessions;
* Has a device with a stable internet connection; and
* Communicates with high school-level English.

Exclusion Criteria:

• Parents with children who have severe behavioral or sensory issues.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-16 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Parental Sense of Competence (PSOC-R) | At the completion of two weeks
  The Parenting Sense of Competence scale (PSOC-R) is a self-report measure that aims to assesses one's perceived efficacy and satisfaction with parenting. 16 items are scored on a scale of 1-6, 1 strongly disagree to 6 strongly agree.
Parent/Caregiver's View of Supporting Children's Play and Playfulness | At the completion of two weeks
  11 items scored on a scale of 0, not agree, to 2, strongly agree, to describe parent's perception of a child's play and joint play.
Strengths and Difficulties Questionnaire (SDQ; Goodman, 1997) | At the completion of two weeks
  Parental self-report assessing a child's behavior, 25 items rated on a scale ranging from 0, not true, to 2, certainly true.

SECONDARY OUTCOMES:
Parent post program open-ended questions | At the completion of two weeks
  A set of three open-ended questions about parents experience and takeaways after participation in the program.
  Can the participants tell the investigators about participant experience with group training? Why do the participants think it worked well and what did not work well for the participants? How do the participants perceive play time with your child/ren now? Has anything changed after the program?
Parent pre program open-ended questions | At enrollment
  A set of three questions regarding parent's expectations of the program.
  The investigators would like to learn more about your thoughts and experiences and will appreciate if the participants could answer the below questions What role does play have in children's development? Do the participants have a designated time that you play with your child? can the participants tell us about it.
  What do the participants expect to gain from these information sessions?

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Fabrizi, PhD OTR/L, Principal Investigator — Associate Professor; AMiya Waldman-Levi, PhD OTR/L, Principal Investigator — Yeshiva University - Professor
Locations (1):
- Little Eagles Learning Center, Fort Myers, Florida, United States

IPD SHARING:
Plan to Share IPD: No
No plans to share participant data.